CLINICAL TRIAL: NCT06240663
Title: A Free-living, Walking-based, Exercise Programme, With Exercise Timed Relative to Breakfast, to Improve Metabolic Health in People Living With Obesity: A Feasibility Study
Brief Title: Walking Before or After Breakfast - Which is Better to Improve Health in Overweight Individuals?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20/SPS021
Record Dates: First submitted 2024-01-03; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Metabolic Disease; Insulin Resistance
MeSH Terms: conditions — Metabolic Diseases; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted (Experimental): Half the participants completed this exercise intervention in the fasted state.
  Interventions: Behavioral: Exercise
- Fed (Experimental): Half the participants completed this exercise intervention in the fed state.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Both groups complete the exercise intervention identically, but one is in the fasted state and one is in the fed state.

SUMMARY:
The aim of this study is to investigate the effectiveness of a home-based walking-based exercise intervention undertaken in the fed or fasted state to improve glycaemic control in overweight and obese individuals. This study will evaluate the adherence and compliance to this "real-world" exercise programme that requires no face-to-face contact with the research team. It is also hypothesised that individuals who exercise before breakfast (fasted) will see greater improvements in glycaemic control than those who exercise after breakfast.

DETAILED DESCRIPTION:
Individuals with a BMI above 28 will be recruited to investigate whether a home-based walking exercise intervention in the fasted or fed state is feasible to implement into real-world situation. Secondary to that, this study will investigate whether a fasted or fed intervention more effective for improving metabolic health. To do this, individuals will provide written consent, and then carry out baseline measures in their own home:

Waist-to-hip ratio and weight: Participants will be provided with a tape measure to measure waist circumference and hip circumference. From this, waist-to-hip ratio will be calculated. Additionally, participants will be asked to use their own scales to provide their weight (if they don't have any they will be provided).

CGM: Participants will receive a continuous blood glucose monitor and be directed over teams how to fit this. One will be worn for two weeks in weeks 0 and 1 and another will be worn for two weeks in weeks 12 and 13.

Diet: Participants will receive a food diary to record their habitual dietary intake for three days (24 hours after the CGM is fitted). During the first week on the intervention they will also be asked to write down what they eat for lunch on the days they exercise.

Fitness test: Participants will receive a polar beat heart rate monitor. They will be asked to complete tthe harvard step test wearing the HR monitor at least 48 hours before they begin the intervention.

Exercise intervention:

Pairs of participants from each group (matched for gender, age, BMI and) will be randomized to undertake 12 weeks of steady walking in either a fasted state (before breakfast each day) or a fed state (after breakfast each day). They will be asked to eat the same breakfast on each day they complete the exercise, whether it is before or after.

Walking sessions will be 4 times per week and will be two continuous sessions (~50% HR max) and two interval sessions (3 minutes at 40% HR max, 3 minutes 80% HR max) monitored by the polar beat app. Participants will initially walk for 30 minute sessions in week 1 and this will increase by 5 minutes each week until they are completing 4x 60 minute sessions per week (see table.1).

A CGM will be in place during week 1 to measure the glycaemic response to exercise. And a second CGM will be inserted at the beginning of week 12 to see the changes in glycaemic control on exercise days and will remain in place for post-intervention CGM monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-60 years
* BMI >28 kg.m-2
* Not currently using any anti-diabetes medication
* Physically inactive (performing less than two 30 min structured exercise sessions per week for the last year)
* Not pregnant or currently breast feeding
* Pre-menopausal or peri-menopausal
* Not currently involved in a weight loss programme or using weight loss medication

Exclusion Criteria:

* Involved in regular exercise (engaged in more than 3 sessions of structured exercise of >30 min per week)
* Currently using anti-diabetes medication (e.g. insulin, metformin)
* Pregnant or breast feeding
* Currently engaged in active weight loss programme or using weight loss medication
* Diagnosed with chronic kidney disease
* Post-menopausal

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Adhearance | Number of exercise sessions are counted. There are 4 exercise sessions prescribed per week for 12 weeks.
  Do individuals complete all the exercise sessions.
Compliance | HR and duration are measured during every exercise session to calculate this. There are 4 exercise sessions prescribed per week for 12 weeks.
  Do participants complete each exercise session as prescribed?

SECONDARY OUTCOMES:
HbA1c | 0 and 12 weeks.
  A Thriva blood sample kit is sent to individuals through the post. t in the post to measure HbA1c, key liver enzymes and cholesterol markers.
Waist circumference | 0 and 12 weeks.
  Participants are sent a tape measure in the post and asked to measure the smallest part of their waist.
Time in Range for Plasma Glucose | Days 0 - 14 and days 77 - 91
  Measured using continuous glucose monitoring
Alanine Transferase | 0 and 12-weeks.
  A Thriva blood sample kit is sent to individuals through the post.
Hip Circumference | 0 and 12-weeks.
  Participants are sent a tape measure in the post and asked to measure the biggest part of their hip.

CONTACTS AND LOCATIONS:
Overall Officials: Sam O Shepherd, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT06240663/Prot_000.pdf
  • Informed Consent Form (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT06240663/ICF_001.pdf